CLINICAL TRIAL: NCT03176394
Title: Efficacy of Bladder Catheters Lubricated With a Biofilm Disruptive Gel, in Reducing Catheter-associated Bacteriuria (CAB) Compared to Standard of Care: A PILOT Clinical Trial
Brief Title: Efficacy of BLASTX in Catheter Associated Bacteriuria Versus Standard of Care (SOC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: trouble with enrollment
Sponsor: Next Science TM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CSP-005
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Urinary Tract Infections
Keywords: Foley, UTI, Biofilm, DNA
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BLASTX Lubricated Catheter (Experimental): Subjects for which catheterization is prescribed will be catheterized with a Foley lubricated with BLASTX. This gel lubricates with the same viscosity as McKesson Jelly and has a biofilm disruptive active ingredient.
  Interventions: Device: BLASTX Gel
- McKesson Jelly Lubricated Catheter (Placebo Comparator): Subjects for which catheterization is prescribed will be catheterized with a Foley lubricated with McKesson Jelly. This jelly lubricates with the same viscosity as BLASTX but has no biofilm disruptive active ingredient.
  Interventions: Device: McKesson Jelly

INTERVENTIONS:
Device: BLASTX Gel — Foley Catheter lubricated with BLASTX Gel
  Arms: BLASTX Lubricated Catheter
Device: McKesson Jelly — Foley Catheter lubricated with McKesson Jelly
  Arms: McKesson Jelly Lubricated Catheter

SUMMARY:
This is a 2-week, single-site, randomized study in adults requiring short-term (≤ 14 days) catheterization. Subjects will be randomized 1:1 to either the biofilm disrupting gel (BLASTX) or SOC (McKesson Jelly) lubricated catheters. Urine and/or catheter DNA analysis will be obtained at catheter insertion, 2, 5, 7 and 14 days after catheterization.

DETAILED DESCRIPTION:
This is a 2-week, single-site, randomized controlled pilot study in adults requiring short-term < 14 days catheterization. Subjects will be randomized 1:1 to either the BLASTX or SOC lubricated catheters.

Urine and catheter DNA analysis will be obtained at catheter insertion, 2 to 3 days after catheterization and at 5, 7 and 14 days if catheterization was indicated for either duration.

Informed consent discussion will be completed, ICF will be signed, prior to any study procedures.

Subjects will be included only if all of the inclusion criteria and none of the exclusion criteria have been met.

After randomization, subjects will be followed, urine samples will be collected at each scheduled visit and the catheters will be collected upon removal.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Absence of symptomatic UTI
3. Absence of upper/lower tract obstructions
4. No known allergies to the study products
5. Willing to comply with all study procedures and available for the duration of the study

Exclusion Criteria:

1. 17 years or younger
2. Symptomatic UTI
3. Presence of upper/lower tract obstructions
4. Known allergic reaction to the study products
5. Unable to provide signed and dated informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Urine microorganisms DNA analysis | Up to 14 days
  Change in microorganisms in the test group compared to the control group.
Catheter microorganisms DNA analysis | Up to 14 days
  Change in microorganisms in the test group compared to the control group.

SECONDARY OUTCOMES:
Incidence of Urinary Tract Infections (UTIs) | 14 days
  Number of instances of clinically symptomatic UTI in the test versus the control group

CONTACTS AND LOCATIONS:
Overall Officials: Susan Greco, MD, Study Director — Next Science
Locations (1):
- American Medical Research Institute, Celebration, Florida, United States

IPD SHARING:
Plan to Share IPD: No